CLINICAL TRIAL: NCT02698033
Title: Follow-Up Protocol For Peanut Allergic Individuals With Documented Objective Clinical Unresponsiveness to a Double-Blind Placebo-Controlled Food Challenge With Peanut Protein
Brief Title: High Threshold Peanut Challenge Study
Acronym: PAID-UP
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Director, Food Allergy Center, Massachusetts General Hospital
Other Study IDs: 2015P001519; 5U19AI095261-02 (NIH)
Record Dates: First submitted 2016-01-29; First posted 2016-03-03 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Peanut Allergy
Keywords: food allergy; peanut; food challenge
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Low dose challenge passed: Individuals who tolerated without dose limiting symptoms the screening food challenge for a parent interventional trial
  Interventions: Drug: Peanut flour; Other: Toasted oat flour

INTERVENTIONS:
Drug: Peanut flour — A Double-blind, placebo-controlled food challenge will consist of two challenges performed on separate days. One challenge will consist of 7 doses of peanut given every 20 minutes in increasing amounts up to a total of 7 grams of whole peanut (4 grams of peanut protein) masked by inclusion in vehicle food. The other challenge will consist of placebo material given similarly.
Other: Toasted oat flour — A Double-blind, placebo-controlled food challenge will consist of two challenges performed on separate days. One challenge will consist of 7 doses of peanut given every 20 minutes in increasing amounts up to a total of 7 grams of whole peanut (4 grams of peanut protein) masked by inclusion in vehicle food. The other challenge will consist of placebo material given similarly.

SUMMARY:
This protocol is designed to better characterize a sub-population of peanut sensitized individuals who may be non-allergic, despite significant sensitization, or who may be allergic, but at high threshold doses. By specifically targeting participants who met the initial screening criteria of the active adult PN OIT study, Protocol 2012p002153 / AADCRC MGH-004 (MGH-004), but failed to react during the pre-treatment 443 mg challenge to peanut, the investigators anticipate that the investigators will identify individuals who have become spontaneously tolerant, despite persistent sensitization. The investigators might also find that clinical sensitivity persists but only with higher thresholds, or that sensitivity has increased (or is variable) since the previous allergen exposure. By repeating DBPCFCs through to a full serving dose (7.4 gram), the investigators will distinguish participants who react only at higher doses from those who were not truly peanut allergic, address whether their sensitivity has changed, and have the opportunity to further investigate their immune response to peanut allergen.

DETAILED DESCRIPTION:
The primary objective of the study is to identify and characterize a sub-population of high-threshold peanut allergic individuals and characterize their immunological phenotype in comparison with the low-threshold peanut allergic individuals enrolled in the adult PN OIT study (NCT01750879).

Clinical Objective:

To evaluate the clinical status of peanut-sensitized individuals previously passing a DBPCFC to 443 mg as being either: non-allergic, stably high-threshold allergic or more clinically reactive on repeat exposure.

ELIGIBILITY:
Inclusion Criteria:

* Failure to react to 443 mg of peanut protein during the DBPCFC1 visit of protocol 2012p002153 / AADCRC MGH-004.
* Males and females of all ethnic/racial groups aged 7-55 years old who are otherwise healthy.
* Willingness to sign consent (or for parent/guardian to sign consent).
* Willingness to sign the assent form, if consent provided by parent/guardian.

Exclusion Criteria:

* History of severe anaphylaxis
* Severe or Moderate asthma
* Poorly controlled asthma
* Diagnosis of other severe or complicating medical problems, including autoimmune or chronic immune inflammatory conditions or gastrointestinal inflammatory conditions
* Inability to cooperate with and/or perform oral food challenge procedures
* Primary Immune Deficiency
* Current use of beta blockers, angiotensin converting enzyme inhibitors, or monoamine oxidase inhibitors
* Women of childbearing potential who are pregnant, planning to become pregnant, or breastfeeding
* Use within the past 6 months of other systemic immunomodulatory treatments
* Clinical signs or symptoms of anemia
* Hematocrit <0.36 for adult females or <0.38 for adult males
* Hematocrit <0.34 for children 7-18 years of age
* Weight <23 kg

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A sub-population of peanut sensitized individuals who may be non-allergic, despite significant sensitization, or who may be allergic, but at high threshold doses.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne G Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peanut Flour: Double Blind Oral food challenge to peanut
  Peanut flour: A food challenge will consist of two challenges performed on separate days. One challenge will consist of 7 doses of peanut given every 20 minutes in increasing amounts up to a total of 7 grams of whole peanut (4 grams of peanut protein) masked by inclusion in vehicle food. The other challenge will consist of placebo material given similarly.
Period: Overall Study
Arm/Group | Peanut Flour
Started | 7
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: A subset of patients screened for NCT01750879 but were not randomized due to threshold reactivity >300 mg peanut protein
Groups:
- Peanut Flour: Double-blind food challenge with peanut flour
  Peanut flour: A Double-blind, placebo-controlled food challenge will consist of two challenges performed on separate days. One challenge will consist of 7 doses of peanut given every 20 minutes in increasing amounts up to a total of 7 grams of whole peanut (4 grams of peanut protein) masked by inclusion in vehicle food. The other challenge will consist of placebo material given similarly.
Arm/Group | Peanut Flour
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Consistency of High Threshold Reactivity
Description: The proportion of high-threshold peanut allergic individuals among participants who previously failed to react to a 443 mg peanut protein challenge in NCT01750879 who also reacted >443 cumulative total dose on repeat challenge
Time Frame: 4 weeks
Population: 1 refused repeat challenge due to other allergic reactivity at time of scheduled procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Flour
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Patient recall of adverse events, with emphasis on accidental ingestion reactions.
Arm/Group | Peanut Flour
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT02698033/Prot_SAP_000.pdf